CLINICAL TRIAL: NCT03929627
Title: Stress in Medical Staff and Controls
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Collaborators: Austrian Federal Ministry of Defence (Unknown)
Responsible Party: Principal Investigator, Michael Sponder, Principal investigator, Medical University of Vienna
Other Study IDs: 1939/2016
Record Dates: First submitted 2017-08-31; First posted 2019-04-29 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Stress
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 - Medical personnell: Group 1 consists of 70 participants belonging to medical staff of the Medical University of Vienna/University Hospital of Vienna and is divided into subgroups consisting of medical technical assistants, nurses, assistant physicians and physicians.
  Interventions: Other: Cortisol awakening response
- Group 2 - Control: Group 2 consists of 70 participants and is recruited from the General non-medical staff of the Austrian Federal Ministry of Defence and Sports, Austrian Armed Forces.
  Interventions: Other: Cortisol awakening response

INTERVENTIONS:
Other: Cortisol awakening response — Cortisol awakening response
  Other Names: Heart rate variability measurement; questionnaires, spiroergometry, laboratory analysis

SUMMARY:
It is expected that medical personnel is exposed to more work-related psychic stress compared to controls and that this burden manifests itself by an increased activity level of the resulting in higher cortisol levels and a decreased HRV. In addition, one is interested in the stress-response/coping strategies of the individuals and believe that regular physical activity might "buffer" the influence of stress on the HPAA-hormones and HRV.

DETAILED DESCRIPTION:
Background Medical personnel is increasingly exposed to psychological stress e.g. caused by work intensification combined with time pressure, fear of job loss, lacking appreciation and/or freedom of decision, causing psychopathological or psychosomatic symptoms involving, inter alia, the cardiovascular system. The aims of the present study are the investigation of the current amount of work-related psychological stress, its perception and underlying reasons, as well as applied recovering strategies (e.g. physical activity) in Austrian health care professionals and in controls.

Material and methods In total, 140 female and male participants (70 participants belong to medical staff; 70 participants belong to non-medical staff) between the ages of 25-65 years will be recruited. The individual stress perception will be evaluated using questionnaires (e.g. Trier Inventory for Chronic Stress, TICS; Brief Symptom Inventory, BSI-18, Short Work Evaluation). 24h salivary cortisol (at 5 time points) and heart rate variability (HRV) measurement will be performed to objectify the influence of stress on the physical body. The physical activity level will be tested by performing a cardiopulmonary exercise test (bicycle spiroergometry).

Expected results From the present study the investigators expects insight into: first, the individual perception of work-related psychological stress among health care professionals compared to the controls; second, the association of occupational stress, HRV and laboratory stress parameters and third, the role of a good physical performance on psychological stress perception.

ELIGIBILITY:
Inclusion Criteria:

* female and male participants aged 25-65 years
* for Group 1: Affiliation to medical staff
* for Group 2: No Affiliation to medical staff

Exclusion Criteria:

* Age <25 or >65 years
* Body weight >130 kg
* Current pregnancy
* Anamnestic current infectious or oncologic disease
* Disability to perform a bicycle stress test
* Atrial fibrillation
* Pace maker/ICD implantation
* Current cortison and/or dexamethasone therapy

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study population consists of 140 female and male participants aged 25-65 years.
  * Group 1 consists of 70 participants belonging to medical staff of the Medical University of Vienna/University Hospital of Vienna and is divided into subgroups consisting of medical technical assistants, nurses, assistant physicians and physicians.
  * Group 2 consists of 70 participants and is recruited from the general staff of the Austrian Federal Ministry of Defence and Sports, Austrian Armed Forces.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-04-30 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Cortisol 1 | Measurement of salivary cortisol right after awakening within 24 hour testing period
  Measurement of salivary cortisol right after awakening
Cortisol 2 | Measurement of salivary cortisol 30 minutes after awakening within 24 hour testing period
  Measurement of salivary cortisol 30 minutes after awakening
Cortisol 3 | Measurement of salivary cortisol at 10 am within 24 hour testing period
  Measurement of salivary cortisol at 10 am
Cortisol 4 | Measurement of salivary cortisol at 4 pm within 24 hour testing period
  Measurement of salivary cortisol at 4 pm
Cortisol 5 | Measurement of salivary cortisol before going to sleep within 24 hour testing period
  Measurement of salivary cortisol before going to sleep

SECONDARY OUTCOMES:
Score of the Work ability Index | once at inclusion
  Comparison of the score of the Work ability Index

OTHER OUTCOMES:
Score of the Effort-Reward Imbalance Questionnaire (ERI) | once at inclusion
  Comparison of the score of the Effort-Reward Imbalance Questionnaire (ERI) by Siegrist
Heart rate variability | once at inclusion over 24 hours, measurement of the parameters every 10 minutes
  Measurement of low frequencies (LF) and high frequencies (HF) by heart rate variability measurement for 24h. The measurement runs for 24h, a median value of the 24h-measurement will be provided.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
Data is available only for the study team